CLINICAL TRIAL: NCT06825013
Title: Bronchodilators and Dynamic Lung Mechanics During Exercise in COPD: Protocol for a Randomised, Placebo-controlled Crossover Trial
Brief Title: Bronchodilators and Lung Mechanics During Exercise in COPD
Acronym: SOUND
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. J. Alberto Neder (Other)
Responsible Party: Sponsor-Investigator, Dr. J. Alberto Neder, Dr. Alberto Neder, Professor, Dept. of Respirology, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOUND STUDY
Record Dates: First submitted 2025-02-03; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: Bronchodilators; Dyspnea; COPD; Exercise; Lung mechanics; Physiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bronchodilator (Active Comparator): Participants will receive a combination short-acting bronchodilator (Salbutamol sulphate (2.5 mg) + ipratropium bromide (0.5 mg)) via nebulizer.
  Interventions: Drug: Bronchodilators inhalation
- Placebo (Placebo Comparator): Participants will receive normal saline via nebulizer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bronchodilators inhalation — Salbutamol sulphate (2.5 mg) + ipratropium bromide (0.5 mg)
  Arms: Bronchodilator
Drug: Placebo — Nebulized saline
  Arms: Placebo

SUMMARY:
Bronchodilators are medications that open the bronchi to help patients with COPD to breathe better. It is still not known exactly how this effect improves shortness of breath in people with COPD. The goal of this clinical trial is to determine whether bronchodilators lower resistance in the smallest airways in the lungs, and whether this will improve the feeling of breathlessness in these patients.

The main questions the investigators attempt to answer are:

* In patients with COPD, does treatment with a short-acting bronchodilator improve small airway resistance during exercise?
* In patients with COPD, does acute treatment with short-acting bronchodilator improve breathlessness and exercise endurance?

The investigators will compare short-acting bronchodilators to placebo (a substance that contains no drug) to see if the bronchodilator medications improve small airway resistance and breathlessness during exercise.

Participants will:

* Visit the research laboratory 3 visits to complete tests of lung function and exercise
* Complete 2 identical visits (Visit 2 and 3), one in which the participant receives bronchodilator and one in which the participant receives placebo.

DETAILED DESCRIPTION:
Small airways disease is a major cause of increased airway resistance and obstruction in chronic obstructive pulmonary disease (COPD). Small airways are those airways beyond generation 8 that are <2 mm in diameter. Due to lung geometry and the mechanism of particle deposition, treatment of small airway disease is challenging and a major clinical concern. Recent advances in respiratory medication delivery devices have purported to improve delivery of medication to the small airways, thus providing better physiologic and symptomatic relief. One such example is Breztri™ Aerosphere©, is a pressurized metered-dose inhaler (pMDI) that delivers triple therapy (long-acting beta-2 agonist, long-acting muscarinic antagonist, and an inhaled corticosteroid), and is currently approved in Canada for patients with COPD. Preliminary evidence has suggested that this product reduced mortality risk and had beneficial effects on exertional dyspnea (shortness of breath), notably in symptomatic patients who have been treated with dry powder inhalers (DPIs). Modeling studies have shown better deposition of drug into the small airways with the pMDI than the DPI; however, it remains unclear whether improved deposition is sufficient to improve small airways function in patients with COPD, and whether these changes result in commensurate improvement in dyspnea and exercise tolerance. Uncovering the mechanisms of dyspnea improvement is a crucial step to provide evidence-based rationale for using pMDI to mitigate the burden of this key patient reported outcome.

Dyspnea during exercise (exertion) in COPD arises when the drive to breathe (neural) is not properly rewarded by the output of the lungs (respiratory mechanics), a phenomenon called "neuromechanical dissociation". In patients with moderate-to-severe COPD, this 'neuromechanical dissociation' is largely a result of impairment in the function of the small airways (airways that are <2mm in diameter) which conspire to induce pulmonary gas trapping and, consequently, increase lung volumes ("hyperinflation"). During exercise when ventilatory demands increase, the reduced time constant for lung emptying (i.e., impaired expiratory time due to increased breathing frequency) leads to acute-on-chronic lung hyperinflation which accelerates attainment of critical inspiratory constraints (i.e., tidal volume expansion is limited), and thus, patients have significantly greater dyspnea and earlier exercise termination. It is reasonable to assume that any inhaled medication for COPD with enhanced access to the small airways could reduce or delay dynamic hyperinflation during exercise and improve a patient's shortness of breath.

MAIN RESEARCH QUESTION In patients with COPD and significant resting lung hyperinflation, does acute treatment with a short-acting bronchodilator (salbutamol sulfate + ipratropium bromide) improve impulse oscillometry derived small airway resistance during cardiopulmonary exercise compared to placebo.

SECONDARY RESEARCH QUESTIONS In patients with COPD and significant resting lung hyperinflation, does acute treatment with short-acting bronchodilator (salbutamol sulfate + ipratropium bromide) improve exertional dyspnea and exercise tolerance during cardiopulmonary exercise compared to placebo. Are improvements in small airway resistance, associated with a reduction in inspiratory neural drive and improved lung mechanics, as measured by diaphragm electromyography (EMGdi).

RESEARCH METHODS Study design: This is a single center, investigator-initiated, prospective, cross over study being conducted over 2-3 weeks.

Study outline:

After giving written informed consent, all participants will be asked to complete 3 visits to the Respiratory Investigation Unit, Kingston General Hospital. Each visit will be conducted at the same time, in the morning, 2 to 7 days apart.

Visit 1 (eligibility assessment): Detailed medical history, physical examination and ECG will be performed. Participants will perform complete pulmonary function testing including spirometry, plethysmography, diffusing capacity for carbon monoxide (DLCO), small airway function assessment (impulse oscillometry (IOS), single-breath and multiple-breath nitrogen washout tests). Participants will complete a symptom-limited incremental cardiopulmonary exercise test (CPET) to determine maximum exercise capacity. PFT and CPET procedures will be conducted according to consensus recommendations.

Visit 2/3 (Constant Work Rate Cardiopulmonary Exercise Test with Placebo or Bronchodilator): Spirometry, body plethysmography, impulse oscillometery, and static and dynamic lung compliance measurements will be performed pre-intervention and 15 minutes post intervention (either dual short-acting bronchodilator (salbutamol sulphate (2.5 mg) + ipratropium bromide (0.5 mg) or a placebo (normal saline)). Participants will then perform a constant work rate tests at 75% peak exercise capacity (determined at V1). Participant will perform exercise on a stationary bicycle while breathing through a mouthpiece with nose clips on, which allows for the breath-by-breath recording of ventilatory and metabolic variables throughout exercise. After approximately 6 minutes of relaxed, baseline breathing, participants will be asked to pedal for 1 minute against no resistance to warm up. The load will then increase to constant work rate (determined at V1), participants will continue to pedal until symptom limitation. Every 2 minutes during exercise, the participant will perform an impulse oscillometery test for assessment of small airways function, followed by an inspiratory capacity maneuver to determine lung volumes. Respiratory discomfort (dyspnea) and leg fatigue will be assessed using the modified Borg 0-10 scale. Vital signs (BP, HR, SpO2) will be monitored throughout each exercise test and during recovery.

Diaphragm EMG and Respiratory Pressure Measurements: At the beginning of Visit 2 and 3, the investigators will apply a topical anesthetic spray to the nasal passages and throat of the participant. A thin catheter (diameter 2 mm) will be inserted by the investigator through the nose down the throat and into the esophagus and top part of stomach. This catheter measures the electric activity (EMG) of the diaphragm, which provides a surrogate measurement of the inspiratory neural drive to breathe. It also measures pressures in the esophagus within the chest as well as in the stomach, which gives useful information about the work of breathing and breathing mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Male or female ≥40-years-of-age
* Current or former smokers with ≥20 pack-year history
* Forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC)<lower limit of normal
* Pre-Post Change of FVC ≥ 10% predicted after 400 mcg inhaled salbutamol
* Functional residual capacity ≥120%predicted and/or the upper limit of normal
* Modified Medical Research Council dyspnea scale ≥ 2
* Clinically stable as defined by no exacerbations in the preceding 6 weeks
* Ability to provide informed consent and perform all study procedures

Exclusion Criteria:

* Major cardiopulmonary diseases other than COPD (asthma, interstitial lung disease, pulmonary hypertension, and congestive heart failure)
* Neuromuscular or musculoskeletal disease
* Use of daytime oxygen or exercise induced O2 desaturation to < 80% on room air;
* Any other disorder that may contribute to exertional dyspnoea and/or exercise intolerance
* Any contraindication to cardiopulmonary exercise testing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Airway resistance | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Primary objective is to measure airway resistance measured by impulse oscillometry at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).

SECONDARY OUTCOMES:
Inspiratory neural drive | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Secondary objective is to measure inspiratory neural drive (IND) by diaphragm activation (EMGdi%max) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Esophageal Pressure (Pes) | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Secondary objective is to measure esophageal pressure (Pes) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Gastric Pressure (Pga) | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Secondary objective is to measure gastric pressure (Pga) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Trans-diaphragmatic Pressure (Pdi) | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Secondary objective is to measure trans-diaphragmatic pressure (Pdi) at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Operating lung volumes | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Secondary objective is to measure inspiratory capacity at isotime (maximum exercise time achieved by all participants) during cardiopulmonary exercise testing (cycle ergometer).
Exertional dyspnea | At 2, 4, 6, 8, and 10 minutes from start of exercise
  Primary objective is to measure perceptual (e.g. intensity of dyspnea) responses at isotime (maximum exercise time achieved by all participants) during a standardized cardiopulmonary exercise testing (cycle ergometer).
Exercise tolerance | Within 10-12 min from start of cardiopulmonary exercise test
  Exercise tolerance will be assessed as the time from start of loaded pedaling to end of loaded exercise.

CONTACTS AND LOCATIONS:
Overall Officials: J Alberto Neder, MD, PhD, Principal Investigator — Queen's University
Locations (1):
- Respiratory Investigation Unit, Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will not be shared until completion of the trial and final analysis. Anonymized data may be made available upon reasonable request after appropriate ethical approval and institutional data sharing agreements
Supporting Information: Study Protocol
Time Frame: Data will not be released until study completion (anticipated January 2027).
Access Criteria: Data will be released on reasonable request after appropriate ethical approval, anonymization, and data sharing agreements to ensure data integrity and participant privacy.